CLINICAL TRIAL: NCT00501878
Title: 2.5% and 10% Phenylephrine for Mydriasis in Diabetic Patients With Darkly Pigmented Irides
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Yosanan Yospaiboon, Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: I50138; HE490619 (Other: Khon Kaen University Ethics Committee)
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus
Keywords: phenylephrine; mydriasis; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Mydriasis | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 2.5% or 10% phenylephrine

SUMMARY:
To compare the clinical efficacy and systemic side effects between 2.5% and 10% phenylephrine for mydriasis in diabetic patient with darkly pigmented irides.

DETAILED DESCRIPTION:
One hundred patients with diabetes from Srinagarind Hospital Eye Clinic were enrolled and randomized into two groups by block randomization. In group I (50 patients), 1% tropicamide combined with 2.5% phenylephrine were administered to dilate pupil whereas 1% tropicamide combined with 10% phenylephrine were used in Group II (50 patients). Pupil diameter, blood pressure and heart rate were measured before and after eye drop instillations.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients

Exclusion Criteria:

* history of intraocular surgery or laser treatment,
* any ocular diseases that might affect pupil size such as glaucoma,uveitis,Horner's syndrome, Adies' pupil,
* history of allergy to any drug used, and
* hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-05; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pupil diameters were measured. | before and after phenylephrine eye drop instillations

SECONDARY OUTCOMES:
blood pressure and heart rate were measured | before and after phenylephrine eye drop instillations

CONTACTS AND LOCATIONS:
Overall Officials: Yosanan Yospaiboon, M.D., Principal Investigator — Khon Kaen University
Locations (1):
- Srinagarind Hospital Eye Clinic, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Result] Suwan-Apichon O, Ratanapakorn T, Panjaphongse R, Sinawat S, Sanguansak T, Yospaiboon Y. 2.5% and 10% phenylephrine for mydriasis in diabetic patients with darkly pigmented irides. J Med Assoc Thai. 2010 Apr;93(4):467-73. PMID 20462091